CLINICAL TRIAL: NCT01133821
Title: Acute Psychotherapy for Bipolar II Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Holly Swartz (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Holly Swartz, Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO08090019; MH084831 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Bipolar Disorder; Depression
Keywords: Bipolar II Disorder; Bipolar II Depression; Psychotherapy; IPSRT; Seroquel; Quetiapine; Placebo; Sugar Pill
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive 20 weeks of an experimental psychotherapy called interpersonal and social rhythm therapy (IPSRT) plus placebo (sugar pill). This condition will be called IPSRT-PLA.
  Interventions: Drug: IPSRT plus placebo (IPSRT-PLA)
- IPSRT plus quetiapine (Experimental): Subjects will receive 20 weeks of an experimental psychotherapy called interpersonal and social rhythm therapy (IPSRT) plus the FDA approved medication quetiapine (Seroquel). This condition will be called IPSRT-QUE.
  Interventions: Drug: IPSRT plus quetiapine

INTERVENTIONS:
Drug: IPSRT plus placebo (IPSRT-PLA) — Subjects will be seen approximately weekly/biweekly during the 20 week acute phase. All subjects will return at weeks 36 and 52 for follow-up assessments to evaluate the enduring effects of treatment.
  The therapist will administer IPSRT and the psychiatrist will administer medication management procedures (quetiapine or placebo).
  Medication Dosing
  The research pharmacy will dispense medication in the following unit-dose packs:
  Dose A (50 mg of QUE or PLA) Dose B (100 mg of QUE or PLA) Dose C (separate packs of 50 mg and 100 mg QUE capsules or PLA) Dose D (200 mg of QUE or PLA) Dose E (separate packs of 50 mg and 200 mg QUE capsules or PLA) Dose F (separate packs of 100mg and 200mg QUE capsules or PLA)
  Other Names: IPSRT-PLA
  Arms: Placebo
Drug: IPSRT plus quetiapine — Subjects will be seen approximately weekly/biweekly during the 20 week acute phase. All subjects will return at weeks 36 and 52 for follow-up assessments to evaluate the enduring effects of treatment.
  The therapist will administer IPSRT and the psychiatrist will administer medication management procedures (quetiapine or placebo).
  Medication Dosing
  The research pharmacy will dispense medication in the following unit-dose packs:
  Dose A (50 mg of QUE or PLA) Dose B (100 mg of QUE or PLA) Dose C (separate packs of 50 mg and 100 mg QUE capsules or PLA) Dose D (200 mg of QUE or PLA) Dose E (separate packs of 50 mg and 200 mg QUE capsules or PLA) Dose F (separate packs of 100mg and 200mg QUE capsules or PLA)
  Other Names: IPSRT-QUE
  Arms: IPSRT plus quetiapine

SUMMARY:
This proposed study is designed to compare the efficacy of interpersonal and social rhythm therapy (IPSRT) alone to IPSRT plus medication as an acute treatment for bipolar II depression. The investigators propose to conduct a randomized, controlled, trial comparing the effects of IPSRT plus pill placebo to IPSRT plus quetiapine on depressive symptoms in individuals suffering from Bipolar II depression. The investigators will also examine the impact of treatment on psychosocial function.

DETAILED DESCRIPTION:
Specifically, we will enroll 160 individuals meeting DSM-IV criteria for BP II disorder, currently depressed, and randomly assign them to 20 weeks of treatment with IPSRT plus placebo (IPSRT-PLA) (N=80) or IPSRT plus quetiapine (IPSRT-QUE) (N=80). We will evaluate potential moderators of response to treatment including circadian phase preference, intercurrent hypomanic symptoms during the index depressive episode, clinical and demographic factors (i.e, number of previous episodes, family history of mood disorders), and prior treatment response to antidepressant medications.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 - 65
* Meets criteria for bipolar II disorder, currently in an episode of major depression, as defined by the DSM-IV (American Psychiatric Association, 1994) and documented by the use of the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I), and by a rating of >15 on the 17-item Hamilton Rating Scale for Depression (HRSD-17)
* Ability and willingness to give informed, written consent.
* Subjects may participate in this study if they are currently taking psychotropic medications at time of informed consent. They will remain in the study (and be randomized) if they still meet eligibility criteria after a one week wash-out period.

Exclusion Criteria:

* Severe or poorly controlled concurrent medical disorders that may cause confounding depressive symptoms (i.e., untreated hypothyroidism or lupus) or require medication(s) that could cause depressive symptoms (i.e., high doses of beta blockers or alpha interferon)
* Meets criteria for one of the following concurrent DSM-IV psychiatric disorders: any psychotic or organic mental disorder, bipolar I disorder, current alcohol or drug dependence, primary obsessive compulsive disorder or primary eating disorders. (primary refers to the diagnosis associated with the most functional impairment); borderline personality disorder; antisocial personality disorder
* Acute suicidal or homicidal ideation or requiring psychiatric hospitalization. Subjects who require inpatient treatment will be excluded (or discontinued) from the study and referred to one of WPIC's inpatient mood disorder units, or, if preferred, to an inpatient facility nearer to the patient's home
* Severe cognitive deficits that would preclude treatment with psychotherapy and/or prevent completion of study questionnaires
* Non-fluent in English. Subjects must be able to speak and understand English because one of the study interventions, IPSRT, is an experimental talk-therapy. This therapy cannot practically be translated.
* Current participation in another form of individual psychotherapy. Concurrent participation in couples therapy, peer support groups (such as Alcoholics Anonymous), or family therapy will be permitted
* Prior lack of response to a trial of at least 12 weeks of IPSRT conducted by a certified therapist
* Prior lack of response to at least 6 weeks of 300 mg of quetiapine
* Currently pregnant or planning to become pregnant during the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Swartz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- WPIC/ Bellefield Towers/Depression and Manic Depression Prevention Program, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Bailey BC, Early TJ, Williams-Sites KE, Dyson B, Swartz HA. Effects of Interpersonal and Social Rhythm Therapy on Suicidal Ideation in Adults With Bipolar II Depression. J Clin Psychiatry. 2025 Sep 29;86(4):24m15768. doi: 10.4088/JCP.24m15768. PMID 41037752
- [Derived] Swartz HA, Rucci P, Thase ME, Wallace M, Carretta E, Celedonia KL, Frank E. Psychotherapy Alone and Combined With Medication as Treatments for Bipolar II Depression: A Randomized Controlled Trial. J Clin Psychiatry. 2018 Mar/Apr;79(2):16m11027. doi: 10.4088/JCP.16m11027. PMID 28703949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: adult outpatients with BD II depression recruited from provider referrals, advertisements, and research registries from 2010-1015
Pre-assignment Details: Participants who met eligibility criteria but were on psychotropic medications at time of informed consent were gradually tapered off medications and re-evaluated to ensure that they still met eligibility criteria following one week off of all medications prior to randomization
Groups:
- Placebo: Subjects will receive 20 weeks of an experimental psychotherapy called interpersonal and social rhythm therapy (IPSRT) plus placebo (sugar pill). This condition will be called IPSRT-PLA.
  IPSRT plus placebo (IPSRT-PLA): Subjects will be seen approximately weekly/biweekly during the 20 week acute phase. All subjects will return at weeks 36 and 52 for follow-up assessments to evaluate the enduring effects of treatment.
  The therapist will administer IPSRT and the psychiatrist will administer medication management procedures (quetiapine or placebo).
  Medication Dosing
  The research pharmacy will dispense medication in the following unit-dose packs:
  Dose A (50 mg of QUE or PLA) Dose B (100 mg of QUE or PLA) Dose C (separate packs of 50 mg and 100 mg QUE capsules or PLA) Dose D (200 mg of QUE or PLA) Dose E (separate packs of 50 mg and 200 mg QUE capsules or PLA) Dose F (separate packs of 100mg and 200mg QUE capsules or PLA)
- IPSRT Plus Quetiapine: Subjects will receive 20 weeks of an experimental psychotherapy called interpersonal and social rhythm therapy (IPSRT) plus the FDA approved medication quetiapine (Seroquel). This condition will be called IPSRT-QUE.
  IPSRT plus quetiapine: Subjects will be seen approximately weekly/biweekly during the 20 week acute phase. All subjects will return at weeks 36 and 52 for follow-up assessments to evaluate the enduring effects of treatment.
  The therapist will administer IPSRT and the psychiatrist will administer medication management procedures (quetiapine or placebo).
  Medication Dosing
  The research pharmacy will dispense medication in the following unit-dose packs:
  Dose A (50 mg of QUE or PLA) Dose B (100 mg of QUE or PLA) Dose C (separate packs of 50 mg and 100 mg QUE capsules or PLA) Dose D (200 mg of QUE or PLA) Dose E (separate packs of 50 mg and 200 mg QUE capsules or PLA) Dose F (separate packs of 100mg and 200mg QUE capsules or PLA)
Period: Overall Study
Arm/Group | Placebo | IPSRT Plus Quetiapine
Started | 45 | 47
Completed | 27 | 28
Not Completed | 18 | 19
Not completed — Lost to Follow-up | 8 | 11
Not completed — Withdrawal by Subject | 8 | 3
Not completed — preferred other treatment | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Refused participation | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | IPSRT Plus Quetiapine | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (11.2) | 30.9 (10.3) | 32.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 19 | 15 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 35 | 31 | 66
  Race: African American | 6 | 10 | 16
  Race: Other | 4 | 6 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 47 | 92

OUTCOME MEASURES:

1. Primary Outcome: Remission
Description: Number of Remitted Participants (defined as 3 consecutive weeks with HRSD-17≤8 and YMRS≤8)
Time Frame: 20 weeks
Population: Intent to treat; patients were assessed weekly
Measure: Count of Participants; unit: Participants
Arm/Group | IPSRT Plus Quetiapine | Placebo
Number analyzed (Participants) | 47 | 45
Participants | 16 | 13
Statistical Analysis 1: Comparison: IPSRT Plus Quetiapine vs Placebo; time effect for HRSD-17; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ)-Short Form
Description: Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ-SF; Total Scores) describes difference in Quality of Life Scores from Baseline to Week 20; The QLESQ-SF is a self-report measure of life satisfaction, with 16 items rated from 1 (very poor) to 5 (very good) to produce a score from 0 to 80 with higher scores indicating better quality of life. In this report, we record change in scores from baseline to follow up
Time Frame: 20 weeks
Population: Analyzed data from participants for whom values were available both at baseline and at twenty weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IPSRT Plus Quetiapine | Placebo
Number analyzed (Participants) | 21 | 26
units on a scale | 10.6 (10.9) | 4.7 (11.4)
Statistical Analysis 1: Comparison: IPSRT Plus Quetiapine vs Placebo; Test type: Superiority; p > 0.05, Regression, Linear; Adjusted for baseline scores

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: Side effects were measured weekly with the Patient Rated Inventory of Side Effects (PRISE), a standardized rating measure of somatic symptoms. Denominators reflect the sample for which the relevant side effect or SAE was measured. SAEs were collected for the total sample; side effects/OAEs were available for a subset of the total sample.
Arm/Group | Placebo | IPSRT Plus Quetiapine
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/47
Other Adverse Events (participants affected / at risk) | 35/44 | 44/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | IPSRT Plus Quetiapine (N=44)
Early Weight Gain (General disorders) | 0 (0) | 2 (2) — (>5% in first month)
Oversedation (General disorders) | 35 (35) | 42 (42) — over-sedation variable was created by combining 3 items from the PRISE (sleeping too much, fatigue, and decreased energy).

LIMITATIONS AND CAVEATS:
Limitations include absence of an inactive psychotherapy comparator, high dropouts, and poor remission rates. Power limitations could potentially leading to Type II errors.Our sample was predominantly white which may limit generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No